CLINICAL TRIAL: NCT04449159
Title: A Randomized, Triple-blind, Placebo-controlled, Parallel Study to Evaluate the Efficacy of Vinh Wellness Collagen on Skin Elasticity, Wrinkles, and Moisturizing Effect
Brief Title: Efficacy of Vinh Wellness Collagen on Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vinh Hoan Corporation (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16ASHV
Record Dates: First submitted 2020-06-19; First posted 2020-06-26 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Skin Manifestations; Skin Abnormalities
MeSH Terms: conditions — Skin Manifestations; Skin Abnormalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Vinh Wellness Collagen (Experimental)
  Interventions: Dietary Supplement: Vinh Wellness Collagen

INTERVENTIONS:
Dietary Supplement: Vinh Wellness Collagen — Vinh Wellness Collagen is hydrolyzed collagen
  Arms: Vinh Wellness Collagen
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The most visible signs of aging are on the skin. As skin gets older it shows a decrease in epidermal thickness, with a flattening of the dermal-epidermal junction. At the same time, loss of elasticity and wrinkle formation begin. The objective of this randomized, triple-blind, placebo-controlled study is to evaluate the efficacy of Vinh Wellness Collagen on skin elasticity, wrinkles, and hydration over 12 weeks.

DETAILED DESCRIPTION:
Skin appearance is known to be influenced by endogenous and environmental factors, including nutrition, hormones, as well as exposure to chemicals, smoking, or ultraviolet radiation. The ability of nutritional supplements to enhance skin characteristics has received increasing attention as the population continues aging. A recent study assessed the correlation between nutrient consumption and skin-aging appearance, including skin wrinkles, dryness, and atrophy, and determined that higher intake of linoleic acid and vitamin C, as well as lower intake of fats and carbohydrates are linked with improved skin appearance. Moreover, clinical trials examining the effects of nutritional supplementation with proteins, vitamins, fatty acids, and trace minerals, have suggested that dietary compounds can modulate skin health and function.

As skin gets older it shows a decrease in epidermal thickness, with a flattening of the dermal-epidermal junction. The dermis is the skin layer directly below the epidermis and has decreases in thickness by about 1% per year throughout the adult lifespan. Structural components of the dermis include collagen, elastic fibers, and extrafibrillar matrix. The cosmetic industry has focused its research on supporting these connective tissue components, as they have been established to repair skin damage (i.e. wounds) and enhance the strength and radiance of the skin.

Collagen is the most abundant protein in mammals and is currently being utilized by a diverse number of industries including nutrition, cosmetic, and biomedical fields. Gelatin, which is used extensively in the food sector, is a hydrolyzed analog of collagen and is an excellent source of protein. A subsequent enzymatic degradation of gelatin results in the generation of collagen hydrolysate (CH), which contains peptides of an average molecular weight of 3-6 kDa. Human bioavailability studies have demonstrated that hydrolyzed collagen peptides are present in the blood within 2 h following oral ingestion of gelatin derived from chicken or fish and are present up to 24 h later.

A double-blind, placebo-controlled trial on 69 women treated with a daily CH treatment or placebo for 8 weeks reported that skin elasticity was significantly improved. Skin moisture and skin evaporation were also enhanced but did not reach statistical significance relative to the placebo group. In addition, other studies have examined the effect of daily ingestion of CH (10 g) or placebo on skin hydration in healthy Japanese women over 2 months and found that there was a gradual improvement in skin water absorption capacity. The objective of this randomized, triple-blind, placebo-controlled study is to evaluate the efficacy of Vinh Wellness Collagen, a CH derived from pangasius skin, on skin elasticity, wrinkles, and hydration over 12 weeks of use.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 45 to 60 years
2. BMI between 20.0-29.9 kg/m2 (±1 kg/m2)
3. Female participant was not of child bearing potential, defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation, or are post-menopausal (natural or surgically with > 1 year since last menstruation)

   OR

   Females of childbearing potential agreed to use a medically approved method of birth control and have a negative urine pregnancy test result. A minimum of 3-months stable dose was required for females on a hormonal birth control. Acceptable methods of birth control included:
   1. Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   2. Double-barrier method
   3. Intrauterine devices
   4. Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   5. Vasectomy of partner (shown successful as per appropriate follow-up)
4. Healthy as determined by laboratory results, medical history, and physical exam
5. No known medical or psychological condition that in the investigator's opinion would interfere with study participation
6. Has given voluntary, written, informed consent to participate in the study
7. Displayed visible signs of natural and photoaging in the face, as assessed through skin condition questionnaire at screening
8. Agreed to avoid prolonged exposure to UV radiation for the duration of the study

Exclusion Criteria:

1. Women who were pregnant, breastfeeding, or planning to become pregnant during the trial
2. Acute or chronic skin disease (i.e. atopic dermatitis, eczema, rosacea, psoriasis) or dermatological disorders (scars, sunburns, moles) near the test sites
3. Topical medications used near the test area within 6 weeks prior to baseline
4. Use of tretinoin, adapalene, tazarotene or other topical medications for the treatment of skin aging near the test site during the 12 weeks preceding baseline
5. Application of topical alpha hydroxyl acids near the test site within 28 days of baseline
6. Use of, or planning to use, systemic corticosteroids within 28 days of baseline or during the study
7. Use of natural health supplements for improving the skin (specifically high concentrations of vitamin A, to be assessed on an individual basis)
8. Planned or unavoidable exposure to intense ultraviolet (UV) radiation during the study (such as sun tanning salons, vacations in a sunny climate or outdoor worker)
9. Botulinum toxin A (Botox) injection treatment near the test sites within 2 years of baseline or plan to receive this treatment during the study
10. Filler injection (collagen, hyaluronic acid, etc.) near the test sites within 2 years of baseline or plan to receive this treatment during the study
11. Tattoos on or near the test area
12. Unstable medical conditions
13. Consumption of more than 2 alcoholic drinks /day
14. Alcohol or drug abuse within 6 months of baseline
15. Tobacco use within 1 year of baseline
16. Use of medical marijuana
17. Participation in clinical research trial within 30 days prior to randomization
18. Allergy or sensitivity to study ingredients or who do not consume fish products (i.e. vegetarians)
19. Participants who were on a low protein diet
20. Cognitively impaired and/or unable to give informed consent
21. Any other condition which in the Investigator's opinion may adversely affect the individual's ability to complete the study or its measures or which may pose significant risk to the individual (e.g. cardiovascular, renal, lung, diabetes, psychiatric illness, bleeding disorders, etc.)

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Cheek skin elasticity | 12 weeks from baseline
  Cheek skin elasticity will be measured using the Cutometer® (MPA 580), which applies the suction method of negative pressure. The skin is drawn into the aperture of the probe using negative pressure, and after a defined time, is released again. The resistance of the skin to the negative pressure (firmness) and its ability to return into its original position (elasticity) are displayed as curves (penetration depth in mm/time) in real time during the analysis.The difference in cheek skin elasticity, measured as Gross skin elasticity (R2), between Vinh Wellness Collagen and placebo supplemented participants after 12 weeks. Cheek skin elasticity will be on a scale of 0-100; 0= no improvement, 100 = great improvement.

SECONDARY OUTCOMES:
Underarm skin elasticity | 12 weeks from baseline
  Underarm elasticity will be measured using the Cutometer® (MPA 580), which applies the suction method of negative pressure. The skin is drawn into the aperture of the probe using negative pressure, and after a defined time, is released again. The resistance of the skin to the negative pressure (firmness) and its ability to return into its original position (elasticity) are displayed as curves (penetration depth in mm/time) in real time during the analysis. The difference in underarm skin elasticity between Vinh Wellness Collagen and placebo supplemented participants after 12 weeks. Underarm skin elasticity will be on a scale of 0-100; 0= no improvement, 100 = great improvement.
Cheek Skin hydration | 12 weeks from baseline
  Cheek skin hydration is evaluated by the Corneometer® (CM 825) using the capacitance method, which is based on the different dielectric constant of water and other substances. Using the corneometer probe, an electric scatter field penetrates ting during the measurement and the dielectricity is determined. The results are stored on the device software as arbitrary units. The difference in cheek skin hydration between Vinh Wellness Collagen and placebo supplemented participants after 12 weeks. Cheek skin hydration will be on a scale of 0-100; 0= no improvement, 100 = great improvement.
Nasolabial wrinkles | 12 weeks from baseliine
  Nasolabial skin wrinkles will be measured by the Modified Fitzpatrick Wrinkle Scale using images acquired by VISIA imaging which utilizes multi-spectral imaging and analysis capture visual information for wrinkles. The difference in nasolabial wrinkles between placebo and Vinh Wellness Collagen participants after 12 weeks of supplementation. The Modified Fitzpatrick Wrinkle Scale (MFWS) is a validated questionnaire that can evaluate skin wrinkle severity. It is on a scale of 0-3; 0 = no wrinkle, 3 = deep wrinkle.
Skin quality using visual analogue scale (VAS) scores | 12 weeks from baseliine
  Skin quality takes account of different measures including skin elasticity, skin hydration, radiance of skin, skin firmness, skin wrinkles and overall feel of skin. Each of these parameters are measured on a scale of 0 - 100; 0 = no improvement. 100 - great improvement. The difference in skin quality VAS scores between placebo and Vinh Wellness Collagen supplemented participants after 12 weeks of supplementation ona scale of 0 - 100; 0 = no improvement, 100 - great improvement.
Net Skin elasticity | Baseline, week 6 and week 12.
  The difference in cheek skin elasticity measured as Net Skin elasticity (R5), between Vinh Wellness Collagen and placebo supplemented participants after 12 weeks. Net skin elasticity is the elastic (immediate stretch) component of the skin without the viscous deformation. Data is represented as the difference between baseline and week 6, baseline and week 12 and between week 6 and week 12. A negative value indicates loss of skin elasticity while a positive number denotes an improved elasticity
Biological elasticity | Baseline, week 6 and week 12.
  This is a measure of skin recovery after deformation. The difference in cheek skin elasticity, measured as biological elasticity (R7), between Vinh Wellness Collagen and placebo supplemented participants after 12 weeks. Data is represented as the difference between baseline and week 6, baseline and week 12 and between week 6 and week 12. A negative value indicates loss of skin elasticity while a positive number denotes an improved elasticity
Viscoelastic recovery (overall elasticity) | 12 weeks from baseliine
  This is a measure of overall skin elasticity. It is calculated using viscous recovery area of the skin relative to the maximum recovery area. Increases in elasticity are considered an improvement.
Systolic and diastolic blood pressure | Baseline, week 6 and week 12.
  Average blood pressure (systolic and diastolic) values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Heart rate | Baseline, week 6 and week 12.
  Average heart rate values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Body weight | Baseline, week 6 and week 12.
  Average body weight values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Body mass index (BMI) | Baseline, week 6 and week 12.
  Average BMI values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Complete blood count (CBC) | Baseline, week 6 and week 12.
  Average CBC values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline and week 6, baseline and week 12 as well as week 6 and week 12.
Aspartate transaminase (AST) | Baseline, week 6 and week 12.
  Average AST values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Alanine transaminase (ALT) | Baseline, week 6 and week 12.
  Average ALT values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Bilirubin | Baseline, week 6 and week 12.
  Average bilirubin values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Sodium ion | Baseline, week 6 and week 12.
  Average sodium ion values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Potassium ion | Baseline, week 6 and week 12.
  Average potassium ion values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Chloride ion | Baseline, week 6 and week 12.
  Average chloride ion values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
Creatinine | Baseline, week 6 and week 12.
  Average creatinine values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.
eGFR | Baseline, week 6 and week 12.
  Average eGFR values for the Vihn Wellness Collagen group will be compared with those of the placebo group using statistical analysis to determine significant difference between the two groups. In addition, within group comparison will be made to determine time-dependent change between baseline versus week 6, baseline versus week 12 as well as week 6 versus week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No